CLINICAL TRIAL: NCT05740098
Title: Financial Incentives for Smoking Cessation Among Disadvantaged Mothers With Young Children
Brief Title: Financial Incentives for Smoking Cessation Among Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Stephen T. Higgins, PhD, Director of the Vermont Center on Behavior and Health and Vice Chair of Department of Psychiatry, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01HD078332 (NIH); R01HD078332 (NIH)
Record Dates: First submitted 2018-12-07; First posted 2023-02-22 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-02

CONDITIONS: Cigarette Smoking
Keywords: Cigarette Smoking; Quit Smoking; Mothers
MeSH Terms: conditions — Cigarette Smoking | interventions — Practice Guidelines as Topic; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Best practices (Experimental): Participants will receive the Five As plus a referral to a quit line.
  Interventions: Behavioral: Best Practices
- Best practices and financial incentives (Experimental): Participants will receive the Five As, a referral to a quit line, and financial incentives contingent on biochemically confirmed smoking abstinence
  Interventions: Behavioral: Best Practices; Behavioral: Financial Incentives
- Best practices, financial incentives, and NRT (Experimental): Participants will receive the Five As, a referral to a quit line, financial incentives contingent on biochemically confirmed smoking abstinence, and nicotine replacement therapy (NRT) provided in the form of both nicotine patches and gum/lozenge for dual therapy.
  Interventions: Behavioral: Best Practices; Behavioral: Financial Incentives; Drug: Nicotine Replacement Therapy

INTERVENTIONS:
Behavioral: Best Practices — Five As plus referral to a quit line
  Other Names: Usual Care
Behavioral: Financial Incentives — Financial incentives provided contingent on biochemically confirmed smoking abstinence. Incentives are in the form of vouchers exchangeable for retail items and available through 12-weeks following quit date.
  Other Names: Contingency Management
  Arms: Best practices and financial incentives; Best practices, financial incentives, and NRT
Drug: Nicotine Replacement Therapy — Nicotine patches and gum/lozenge provided together for dual therapy
  Other Names: NRT
  Arms: Best practices, financial incentives, and NRT

SUMMARY:
Investigators will examine whether adding financial incentives and nicotine replacement dual therapy to current best practices for smoking cessation (i.e. referral to counseling using a telephone quit line) increases cessation rates in mothers and reduces second-hand smoke exposure in children. While perhaps more expensive upfront compared to best practices alone, the investigators hypothesize that this treatment approach will be a more cost-effective cessation intervention.

DETAILED DESCRIPTION:
Smoking prevalence among disadvantaged mothers remains at strikingly high levels (40-60%). Disadvantaged women are more likely to begin smoking at an earlier age, be heavier smokers, be nicotine dependent, and fail in their efforts to quit smoking (Kandel et al., 2009). These women and their children also suffer higher rates of smoking-related adverse health consequences.

Despite widespread knowledge of the harmful effects of secondhand smoke exposure (SHSe), estimates are that 85% of children from low-income U.S. families experience chronic exposure. Children exposed to SHS are at increased risk for numerous serious health problems, including sudden infant death syndrome, more severe asthma, lower respiratory infections, and chronic middle ear disease, and maternal smoking is a particularly significant contributor to this increased morbidity and mortality. SHSe is also a substantial economic burden on the U.S. healthcare system, being estimated to increase direct medical and life-lost costs by > $5 billion annually.

Interventions developed to reduce children's SHSe have aimed to (1) decrease parental smoking around their children, (2) increase parental smoking cessation, or (3) both. Since smoking by a child's mother is a particularly significant contributor to SHSe, interventions have typically targeted smoking mothers. Regarding efforts to decrease smoking around children, studies testing relatively low-intensity interventions (e.g., written materials, brief advice) have failed to change exposure levels, while those testing more intensive interventions have had more success decreasing children's SHSe, with at least some instances of biochemically-verified changes.

Clearly, more effective smoking-cessation interventions for mothers are needed to meet the public health priority of reducing SHSe among children. The investigators recognize that maternal smoking cessation will not eliminate SHSe among children since many (~40%) live with more than one smoker. However, the evidence is clear that smoking mothers are the primary contributors to their children's SHSe, making them the obvious first target. The overarching goal of this project is to develop an efficacious, cost-effective incentive-based smoking cessation intervention that is combined with state-of-the-art smoking-cessation pharmacotherapy practices to optimize outcomes.

Participants will be 250 mothers (10 pilot and 80 per treatment condition) recruited from our university-affiliated hospital's pediatric practice, other pediatric and family medicine practices throughout the county in which our clinic is located, local offices for Women, Infants, and Children (WIC), and other recruitment strategies (e.g., ads on Facebook). Participants will be randomly assigned to one of three treatment conditions: (1) usual care for smoking cessation and protecting children from SHSe, (2) usual care combined with incentives for objectively verified smoking abstinence, and (3) usual care combined with incentives and pharmacotherapy using innovative procedures to enhance its efficacy.

The investigators believe combining pharmacotherapies with incentives could be an effective strategy for surmounting adherence problems in this population by assuring that women have regular contact with clinic staff and thereby providing staff opportunities to problem-solve obstacles that may have arisen around adherence or side effects and to regularly underscore the importance and potential benefits of using the medications as prescribed.

The investigators hypothesize that each of the interventions with incentives will increase smoking abstinence compared to usual care alone, but that the largest magnitude and most cost-effective treatment effects will be achieved by combining incentives with pharmacotherapy. They also hypothesize that (a) both incentives interventions will decrease child cotinine levels significantly more than usual care alone and (b) that SHSe levels will be significantly lower among children of abstainers than smokers.

Taken together, developing efficacious and cost-effective interventions to increase smoking cessation interventions among disadvantaged mothers and reducing SHSe among their children is an important U.S. public health priority. The financial incentives model is effective with other treatment-recalcitrant populations and we believe has the potential to meet this important public-health challenge. Behavioral-economic theory suggests that the efficacy of the cessation intervention is at least in part attributable to providing smaller, more immediate incentives for success that act to bridge the temporal delay to the larger naturalistic rewards of improved health outcomes for mother and child. The investigators will continue to investigate the behavioral-economic processes involved in smoking among disadvantaged women and in individual differences in treatment response. Lastly, there is rapidly growing interest in the use of incentives to promote healthy behavior change in disadvantaged populations. The proposed project and others like it will be important to assuring that the necessary scientific knowledge is available to support that effort.

ELIGIBILITY:
Inclusion Criteria:

* Expresses interest in quitting smoking
* Express willingness to initiate NRT
* Mother is ≥ 18 years of age
* Self-reported smoking ≥ 10 cigarettes per day for ≥ 1 year, biochemically verified
* Mother has a child < 12 years of age
* Child resides with mother full-time
* Not currently using any other tobacco cessation medications (e.g. Chantix) or NRT, or willing to stop use prior to participation in the study
* Lives in Chittenden County, Vermont or surrounding counties
* Plans on remaining in the geographical area for the next 12 months
* English-speaking
* Willing to let child participate in the study

Exclusion Criteria:

* Failing to meet any of the above criteria
* Has medical contraindications to NRT products
* Meeting Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for moderate or severe alcohol or drug dependence other than nicotine in the prior 12 months (those on opioid substitution therapy are allowed)
* Current/past psychotic disorder
* Being suicidal
* Currently pregnant or trying to become pregnant in the next 12 months
* Incarceration
* Refusal to participate in study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T Higgins, PhD, Study Director — University of Vermont
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Higgins ST, Plucinski S, Orr E, Nighbor TD, Coleman SRM, Skelly J, DeSarno M, Bunn J. Randomized clinical trial examining financial incentives for smoking cessation among mothers of young children and possible impacts on child secondhand smoke exposure. Prev Med. 2023 Nov;176:107651. doi: 10.1016/j.ypmed.2023.107651. Epub 2023 Jul 30. PMID 37527730

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Best Practices | Best Practices and Financial Incentives | Best Practices, Financial Incentives, and NRT
Started | 68 | 63 | 67
Completed | 42 | 46 | 46
Not Completed | 26 | 17 | 21
Not completed — Lost to Follow-up | 26 | 17 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Best Practices | Best Practices and Financial Incentives | Best Practices, Financial Incentives, and NRT | Total
Number analyzed (Participants) | 68 | 63 | 67 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.95 (5.86) | 31.82 (6.18) | 32.88 (6.50) | 32.56 (6.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 63 | 67 | 198
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 60 | 57 | 60 | 177
  Other | 8 | 6 | 7 | 21
Region of Enrollment [Number; unit: participants]
  United States | 68 | 63 | 67 | 198
Maternal smoking status [Count of Participants; unit: Participants]
  Smoking | 68 | 63 | 67 | 198
  non-smoker | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence Smoking Abstinence Levels
Description: Point prevalence abstinence will be defined as self-report of no smoking in the past 7 days, not even a puff, with biochemical verification via breath carbon monoxide (CO) and urine cotinine. Abstinence at the 12-week (end of treatment) and 24-week assessment will be compared between the three treatment arms.
Time Frame: Collected once per woman at approximately 12- and 24- weeks following quit date in each of the three smoking arms
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practices | Best Practices and Financial Incentives | Best Practices, Financial Incentives, and NRT
Number analyzed (Participants) | 68 | 63 | 67
Participants
  12 weeks | 4 | 22 | 18
  24 weeks | 6 | 14 | 12
Statistical Analysis 1: Comparison: Best Practices vs Best Practices and Financial Incentives; Analysis tested for significant main effects of treatment condition on 7-day point prevalence abstinence at 12- and 24-week assessments; Test type: Superiority; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 5.378, 95% CI 2-sided [2.278 to 12.689]
Statistical Analysis 2: Comparison: Best Practices vs Best Practices, Financial Incentives, and NRT; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.003, Mixed Models Analysis; Odds Ratio (OR) = 3.668, 95% CI 2-sided [1.538 to 8.747]
Statistical Analysis 3: Comparison: Best Practices and Financial Incentives vs Best Practices, Financial Incentives, and NRT; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.256, Mixed Models Analysis; Odds Ratio (OR) = 0.682, 95% CI 2-sided [0.352 to 1.321]
Statistical Analysis 4: Comparison: Best Practices vs Best Practices and Financial Incentives vs Best Practices, Financial Incentives, and NRT; Analysis tested for significant main effect of time on 7-day point prevalence abstinence at 12- and 24-week assessments; Test type: Superiority; p < 0.001, Mixed Models Analysis

2. Primary Outcome: Objective Measure of Child Secondhand Smoke Exposure (SHSe)
Description: SHSe will be defined as the level of cotinine measured in the urine of the youngest child at baseline, 6-, 12-, and 24-weeks following the mother's quit date. SHSe outcomes will be compared between the three treatment arms and between children of abstainers versus smokers independent of treatment condition. We hypothesize being able to detect greater reductions from baseline levels in the incentives compared to Best Practices treatment conditions and among abstainers compared to smokers. We report main effects of treatment condition as geometric means (+/- SEM) collapsed across the three assessment times for each treatment condition controlling for baseline values.
Time Frame: Collected twice per child at baseline, and once at approximately 6-, 12- and 24-weeks following quit date
Population: This analysis is based on only children who submitted a baseline and at least one valid urine specimen between Weeks 6-24. Note that numbers in the Overall Participant Flow pertains to mothers while those shown in this section pertain to children.
Measure: Geometric Least Squares Mean (Standard Error); unit: ng/ml
Arm/Group | Best Practices | Best Practices and Financial Incentives | Best Practices, Financial Incentives, and NRT
Number analyzed (Participants) | 52 | 47 | 51
ng/ml | 3.53 (0.96) | 3.48 (0.92) | 8.49 (2.22)
Statistical Analysis 1: Comparison: Best Practices vs Best Practices and Financial Incentives; Analysis tested for significant main effect of treatment condition on Child Urine Cotinine; Test type: Superiority; p = 0.287, Mixed Models Analysis; Mean Difference (Final Values) = 0.39, Standard Error of Mean 0.365
Statistical Analysis 2: Comparison: Best Practices vs Best Practices, Financial Incentives, and NRT; Analysis tested for significant main effect of treatment condition on Child Urine Cotinine; Test type: Superiority; p = 0.108, Mixed Models Analysis; Mean Difference (Final Values) = -0.597, Standard Error of Mean 0.369
Statistical Analysis 3: Comparison: Best Practices and Financial Incentives vs Best Practices, Financial Incentives, and NRT; Analysis tested for significant main effect of treatment condition on Child Urine Cotinine; Test type: Superiority; p = 0.007, Mixed Models Analysis; Mean Difference (Final Values) = -0.987, Standard Error of Mean 0.361
Statistical Analysis 4: Comparison: Best Practices vs Best Practices and Financial Incentives vs Best Practices, Financial Incentives, and NRT; Analysis tested for significant main effect of time on Child Urine Cotinine; Test type: Superiority; p = 0.878, Mixed Models Analysis

3. Secondary Outcome: Continuous Abstinence
Description: Continuous abstinence will be defined as self-report of no smoking in the past 7 days at each time point, not even a puff, with biochemical verification via breath CO and urine cotinine. Continuous abstinence from quit date through 24 week assessment will be compared between the three treatment arms.
Time Frame: 24 weeks following quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practices | Best Practices and Financial Incentives | Best Practices, Financial Incentives, and NRT
Number analyzed (Participants) | 68 | 63 | 67
Participants | 3 | 12 | 10
Statistical Analysis 1: Comparison: Best Practices vs Best Practices and Financial Incentives; Analysis tested for significant main effect of treatment condition on continuous abstinence at 24 weeks following quit date; Test type: Superiority; p = 0.009, Chi-squared; Degrees of freedom = 1; Chi-Square Test Statistic = 6.909
Statistical Analysis 2: Comparison: Best Practices vs Best Practices, Financial Incentives, and NRT; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.038, Chi-squared; Degrees of freedom = 1; Chi-Square Test Statistic = 4.287
Statistical Analysis 3: Comparison: Best Practices and Financial Incentives vs Best Practices, Financial Incentives, and NRT; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.531, Chi-squared; Degrees of freedom = 1; Chi-Square Test Statistic = 0.392

4. Secondary Outcome: 7-day Point Prevalence Abstinence at 48-week Follow-up Assessment
Description: Point prevalence abstinence will be defined as self-report of no smoking in the past 7 days, not even a puff, with biochemical verification via breath CO and urine cotinine. We will use this data to estimate relapse rates across treatment arms and for use in comparing SHSe levels in children of abstainers versus smokers.
Time Frame: 48 weeks following quit date
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practices | Best Practices and Financial Incentives | Best Practices, Financial Incentives, and NRT
Number analyzed (Participants) | 68 | 63 | 67
Participants | 5 | 11 | 6
Statistical Analysis 1: Comparison: Best Practices vs Best Practices and Financial Incentives vs Best Practices, Financial Incentives, and NRT; Analysis tested for significant main effect of treatment condition on 7-day point prevalence abstinence at 48-week follow-up; Test type: Superiority; p = 0.145, Chi-squared; Degrees of freedom = 2; Chi-Square Test Statistic = 3.859

5. Secondary Outcome: Smoking Abstinence
Description: Biochemically-verified 7-day point-prevalence smoking abstinence.
Time Frame: Assessed once per woman at 6-, 12-, 24-, and 48-weeks following quit date.
Population: Participants who completed a valid baseline delay-discounting assessment. Six participants did not have a valid assessment making total N 192 rather than 198 participants. Analyses tested for interactions of treatment and delay discounting. If there is a significant interaction (P < 0.05) of treatment condition and baseline delay discounting, we report results separately by treatment condition. In the absence of significant interactions, we collapse results across treatment conditions.
Measure: Count of Participants; unit: Participants
Groups:
- Collapsing Participants Across Treatment Conditions: We examined association between baseline temporal discounting and abstinence achieved at follow-up assessments collapsing participants across treatment conditions.
Arm/Group | Collapsing Participants Across Treatment Conditions
Number analyzed (Participants) | 192
Participants
  # abstinent 6-wks | 49
  # abstinent 12-wks | 44
  # abstinent 24-wks | 32
  # abstinent 48-wks | 22
Statistical Analysis 1: Comparison: Collapsing Participants Across Treatment Conditions; Analysis tested for significant main effect of baseline temporal discounting on point-prevalence abstinence at 6-weeks following quit date adjusting for treatment condition; Test type: Superiority; p = 0.228, Regression, Logistic; Wald Chi-Square Test Statistic = 1.454
Statistical Analysis 2: Comparison: Collapsing Participants Across Treatment Conditions; Analysis tested for significant main effect of baseline temporal discounting on point-prevalence abstinence at 12-weeks following quit date adjusting for treatment condition; Test type: Superiority; p = 0.10, Regression, Logistic; Wald Chi-Square Test Statistic = 2.70
Statistical Analysis 3: Comparison: Collapsing Participants Across Treatment Conditions; Analysis tested for significant main effect of baseline temporal discounting on point-prevalence abstinence at 24-weeks following quit date adjusting for treatment condition; Test type: Superiority; p = 0.074, Regression, Logistic; Wald Chi-Square Test Statistic = 3.202
Statistical Analysis 4: Comparison: Collapsing Participants Across Treatment Conditions; Analysis tested for significant main effect of baseline temporal discounting on point-prevalence abstinence at 48-weeks following quit date adjusting for treatment condition; Test type: Superiority; p = 0.484, Regression, Logistic; Wald Chi-Square Test Statistic = 0.491

6. Secondary Outcome: Smoking Abstinence
Description: Biochemically-verified 7-day point-prevalence smoking abstinence.
Time Frame: Collected once per woman at baseline, 6-, 12-, 24-, and 48-weeks following quit date.
Population: Participants who completed a valid baseline Cigarette-Purchase-Task (CPT) assessment. Ten participants did not have a valid assessment making total N 188 rather than 198 participants. Analyses tested for interactions of treatment and CPT Latent Factors. If there is a significant interaction (P < 0.05) of treatment condition and CPT Latent Factors, we report results separately by treatment condition. In the absence of significant interactions, we collapse results across treatment conditions.
Measure: Count of Participants; unit: Participants
Groups:
- Collapsing Participants Across Treatment Conditions: We examined association between baseline price sensitivity (latent factors Amplitude and Persistence) and abstinence achieved at follow-up assessments collapsing participants across treatment conditions.
Arm/Group | Collapsing Participants Across Treatment Conditions
Number analyzed (Participants) | 188
Participants
  # abstinent 6-wks | 49
  # abstinent 12-wks | 44
  # abstinent 24-wks | 32
  # abstinent 48-wks | 22
Statistical Analysis 1: Comparison: Collapsing Participants Across Treatment Conditions; The analysis tested for significant association between baseline price sensitivity (latent factor Amplitude) and abstinence at 6-weeks following quit date; Test type: Superiority; p = 0.302, Regression, Logistic; Wald Chi-Square Test Statistic = 1.063
Statistical Analysis 2: Comparison: Collapsing Participants Across Treatment Conditions; The analysis tested for significant association between baseline price sensitivity (latent factor Amplitude) and abstinence at 12-weeks following quit date; Test type: Superiority; p = 0.375, Regression, Logistic; Wald Chi-Square Test Statistic = 0.788
Statistical Analysis 3: Comparison: Collapsing Participants Across Treatment Conditions; The analysis tested for significant association between baseline price sensitivity (latent factor Amplitude) and abstinence at 24-weeks following quit date; Test type: Superiority; p = 0.777, Regression, Logistic; Wald Chi-Square Test Statistic = 0.080
Statistical Analysis 4: Comparison: Collapsing Participants Across Treatment Conditions; The analysis tested for significant association between baseline price sensitivity (latent factor Amplitude) and abstinence at 48-weeks following quit date; Test type: Superiority; p = 0.937, Regression, Logistic; Wald Chi-Square Test Statistic = 0.006
Statistical Analysis 5: Comparison: Collapsing Participants Across Treatment Conditions; The analysis tested for significant association between baseline price sensitivity (latent factor Persistence) and abstinence at 6-weeks following quit date; Test type: Superiority; p = 0.678, Regression, Logistic; Wald Chi-Square Test Statistic = 0.172
Statistical Analysis 6: Comparison: Collapsing Participants Across Treatment Conditions; The analysis tested for significant interaction between baseline price sensitivity (latent factor Persistence) and treatment condition for 6-week abstinence outcome; Test type: Superiority; p = 0.018, Regression, Logistic; Wald Chi-Square Test Statistic = 7.99
Statistical Analysis 7: Comparison: Collapsing Participants Across Treatment Conditions; The analysis tested for significant association between baseline price sensitivity (latent factor Persistence) and abstinence at 12-weeks following quit date; Test type: Superiority; p = 0.674, Regression, Logistic; Wald Chi-Square Test Statistic = 0.177
Statistical Analysis 8: Comparison: Collapsing Participants Across Treatment Conditions; The analysis tested for significant association between baseline price sensitivity (latent factor Persistence) and abstinence at 24-weeks following quit date; Test type: Superiority; p = 0.422, Regression, Logistic; Wald Chi-Square Test Statistic = 0.646
Statistical Analysis 9: Comparison: Collapsing Participants Across Treatment Conditions; The analysis tested for significant association between baseline price sensitivity (latent factor Persistence) and abstinence at 48-weeks following quit date; Test type: Superiority; p = 0.846, Regression, Logistic; Wald Chi-Square Test Statistic = 0.038

7. Other Pre Specified Outcome: Number of Outpatient Child Visits to Healthcare Center.
Description: Number of outpatient child visits will be compared between the three treatment arms and between abstainers versus smokers, independent of treatment condition.
Time Frame: 48 weeks following quit date.
Population: Data collection on this outcome was to occur following completion of data collection on treatment outcomes. The COVID pandemic prevented data collection on this outcome.
Groups:
- Treatment Condition: Data not collected in any treatment condition.
Arm/Group | Treatment Condition
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Number of Inpatient Child Visits to Healthcare Center.
Description: Number of inpatient child visits will be compared between the three treatment arms and between abstainers versus smokers, independent of treatment condition.
Time Frame: 48 weeks following quit date.
Population: as for outcome 7
Arm/Group | Treatment Condition
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Number of Times Child Received Prescription Medications.
Description: Number of times child received prescription medications will be compared between the three treatment arms and between abstainers versus smokers, independent of treatment condition.
Time Frame: 48 weeks following quit date.
Population: as for outcome 7
Arm/Group | Treatment Condition
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Cost-effectiveness Analysis
Description: Cost-effectiveness will include the cost of each intervention, measured by the Brief Drug Abuse Treatment Cost Analysis Program (Brief-DATCAP) and the economic cost of treatment (fixed costs based upon proportion of time and/or space utilized by the program). Estimated treatment costs will be combined with estimated child healthcare utilization costs to represent total costs per treatment condition. Treatment costs will be compared across the three treatment arms.
Time Frame: Study entry through 48 weeks following quit date.
Population: Cost-effectiveness analysis was not conducted because data collection on necessary outcomes was not completed due to the COVID pandemic.
Arm/Group | Treatment Condition
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected across 48 weeks following study entry for each participant.
Arm/Group | Best Practices | Best Practices and Financial Incentives | Best Practices, Financial Incentives, and NRT
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/63 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/68 | 1/63 | 0/67
Other Adverse Events (participants affected / at risk) | 0/68 | 0/63 | 0/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Best Practices (N=68) | Best Practices and Financial Incentives (N=63) | Best Practices, Financial Incentives, and NRT (N=67)
Serious Adverse event (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Participant obtained transdermal nicotine replacement therapy from her primary care physician. She used greater than recommended dose of transdermal nicotine plus an e-cigarette resulting in gastric upset and treatment in Emergency Department.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT05740098/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT05740098/SAP_001.pdf